CLINICAL TRIAL: NCT06076018
Title: The Contribution of Intrathecal Morphine Administration to Postoperative Patient Satisfaction During Cesarean Delivery
Acronym: ITM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilke Tamdogan, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: drilketamdogan
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Cesarean Section; Intrathecal Morphine; Quality of Recovery 40
Keywords: Quality of Recovery 40; intrathecal morphine; cesarean section

STUDY DESIGN:
Intervention Model Description: In the study planned as a randomized clinical study, patients who use and do not use intrathecal morphine will be assigned to 2 groups, 30 people in each group, by the sealed envelope method. Patients, surgeons, and physicians who will perform postoperative evaluation and fill out the questionnaire will be blinded to the randomization of the groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrathecal morphine (Active Comparator): In spinal anesthesia, 12 mg hyperbaric bupivacaine and 20 mcg fentanyl, 120 mcg intrathecal morphine (ITM) will be administered intrathecally.
  Interventions: Drug: Group morphine
- intrathecal fentanyl (Placebo Comparator): Intrathecal 12 mg hyperbaric bupivacaine and 20 mcg fentanyl in spinal anesthesia, ITM will not be applied
  Interventions: Other: Group placebo

INTERVENTIONS:
Drug: Group morphine — Spinal anesthesia will be applied to patients in a sitting position, with a midline approach, after aseptic conditions have been achieved. A 25 gauge pencil point spinal needle will be placed in the L3-4 or L4-5 space. Upon aspiration of clear cerebrospinal fluid (CSF), 12 mg hyperbaric bupivacaine and 20 mcg fentanyl will be administered intrathecally, and 120 mcg intrathecal morphine (ITM) will be administered to the morphine group. the 24th postoperative hour, all patients will be visited in the ward and the QoR-40 (Quality of Recovery-40) patient satisfaction recovery quality scale, scored between 40-200, will be filled out.
  Other Names: intrathecal morphine
  Arms: intrathecal morphine
Other: Group placebo — Spinal anesthesia will be applied to patients in a sitting position, with a midline approach, after aseptic conditions have been achieved. A 25 gauge pencil point spinal needle will be placed in the L3-4 or L4-5 space. Upon aspiration of clear cerebrospinal fluid (CSF), 12 mg hyperbaric bupivacaine and 20 mcg fentanyl will be administered intrathecally. the 24th postoperative hour, all patients will be visited in the ward and the QoR-40 (Quality of Recovery-40) patient satisfaction recovery quality scale, scored between 40-200, will be filled out.
  Other Names: control
  Arms: intrathecal fentanyl

SUMMARY:
Evaluating the contribution of intrathecal morphine administration to postoperative patient satisfaction during cesarean delivery with the QoR-40 (Quality of Recovery 40) patient satisfaction compilation quality scale, scored between 40-200, and demonstrating the difference in the global QoR-40 score.

DETAILED DESCRIPTION:
All patients, whose consent was obtained, were monitored for standard noninvasive blood pressure, heart rate (HR), electrocardiogram (ECG) findings, and peripheral oxygen saturation (SpO2) in the operating room.

Patients were evaluated for side effects such as pain, nausea-vomiting, itching, sedation score, and respiratory depression (defined as respiratory rate <10/min or SpO2<93%) for 24 hours postoperatively. Evaluations were made at the 2nd, 4th, 6th, 8th, 12th and 24th hours postoperatively. Pain assessment was made with the 'Numeric Rating Scale' (NRS) (0-10, 0 = no pain and 10 = worst pain imaginable), sedation assessment was made with the 'Ramsey Sedation Scale'. Nausea was evaluated as present or absent (0:absent, 1:present) and itching 'Verbal Descriptive Scale' (0: no itching, 1: was evaluated using mild, 2: moderate, 3: severe, 4: very severe).

At the 24th postoperative hour, all patients were visited in the ward and the QoR-40 (Quality of Recovery-40) patient satisfaction compilation quality scale, scored between 40-200, was filled out. The QoR-40 questionnaire is a self-rating questionnaire used to evaluate the quality of postoperative recovery and health status of patients in the early postoperative stages. For the first time, Myles et al. () in 2000 and was proven to be a valid test in Turkey by Karaman S. et al. in 2014. QoR-40 was used to evaluate the pain levels, physical and emotional status of patients; emotional state (n = 9), comfort ( It consists of five sections and 40 questions: n = 12), patient support (n = 7), physical independence (n = 5), and pain (n = 7). Each question is scored on a five-point Likert scale ranging from 1 to 5. The total score ranges from 40 (worst build quality) to 200 (best build quality).

This widely used survey has been successfully applied to populations with cultural and physical differences in many different countries. QoR-40 studies conducted after a wide variety of anesthesia and surgical techniques reveal how wide the field of use of the test is. As a result of all this, the researchers reported that the test was safe and applicable.

Maternal characteristics such as age, weight, height, gestational age, gravidity, parity, number of previous cesarean births and procedure time, and tubal ligation were recorded. Newborn characteristics were collected, including weight and Apgar scores

ELIGIBILITY:
Inclusion Criteria:

* Between 18-40 years old,
* ASA physical status 2
* Patients who will give birth by elective cesarean section

Exclusion Criteria:

* Those who do not accept regional anesthesia,
* Pregnant women who have problems where spinal anesthesia is contraindicated, such as infection at the injection site, coagulopathy, bleeding diathesis, severe hypovolemia, increase in intracranial pressure, severe aortic stenosis, severe mitral stenosis,
* Patients with a history of allergy to any drug included in the study protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Difference in QoR-40 score at 24th postoperative hour | Postoperative Day 1
  Evaluation of the contribution of intrathecal morphine application to postoperative patient satisfaction during cesarean delivery with the QoR-40 (Quality of Recovery 40) patient satisfaction compilation quality scale scored between 40-200 and the difference in the global QoR-40 score

SECONDARY OUTCOMES:
Post-operative acute pain | Postoperative Day 1
  Pain status at rest and while activity (coughing and walking) was assessed by NRS scores at 2, 4, 6, 8, 12 and 24 hours after surgery. The NRS is an 11-point numeric scale which ranges from 0 to 10 at rest and during activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Karaman S, Arici S, Dogru S, Karaman T, Tapar H, Kaya Z, Suren M, Gurler Balta M. Validation of the Turkish version of the Quality of Recovery-40 questionnaire. Health Qual Life Outcomes. 2014 Jan 15;12:8. doi: 10.1186/1477-7525-12-8. PMID 24428925